CLINICAL TRIAL: NCT04417998
Title: Improving PET Image Quality and Quantification by Using Motion Correction, Parametric Imaging and MAP Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bradley Kemp, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-010591
Record Dates: First submitted 2020-04-14; First posted 2020-06-05 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Brain Imaging; Whole Body Imaging
Keywords: Brain Imaging; Whole Body Imaging
MeSH Terms: interventions — Fluorodeoxyglucose F18; 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study. Aim 1 involves the prospective data collection of subjects who are already enrolled in Mayo Clinic Rochester research study 08-005553 (PI: Dr Val Lowe) and are scheduled to be scanned on the Siemens Biograph Vision 600 PET/CT system (hereafter referred to as the V600-R1) in the PET/CT Molecular Imaging Research Center on Charlton 6 of Mayo Clinic Rochester. Aim 2 involves the prospective data collection of subjects undergoing brain or whole body oncologic PET/CT scans on the V600-R1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Motion Correction (Active Comparator): Aim 1 involves the prospective data collection of subjects who are already enrolled in Mayo Clinic Rochester research study 08-005553 (PI: Dr Val Lowe) and are scheduled to be scanned on the Siemens Biograph Vision 600 PET/CT system (hereafter referred to as the V600-R1) in the PET/CT Molecular Imaging Research Center on Charlton 6 of Mayo Clinic Rochester. The purpose of this arm is to evaluate the effectiveness of motion correction software.
  Interventions: Device: Siemens E7 Reconstruction Tool
- Parametric Imaging (Active Comparator): Aim 2 involves the prospective data collection of subjects undergoing brain or whole body oncologic PET/CT scans on the V600-R1. The purpose of this arm is to evaluate the data acquisition and image processing workflow.
  Interventions: Drug: 18F-FDG; Drug: 18F-AV1451

INTERVENTIONS:
Drug: 18F-FDG — A cohort of participants in Aim 2 will undergo a 18F-FDG PET/CT scan. This scan is done with a radiotracer called 18F-fluorodeoxyglucose (FDG). FDG looks at cellular activity.
  Other Names: FDG
  Arms: Parametric Imaging
Drug: 18F-AV1451 — A cohort of participants in Aim 2 will undergo a 18F-AV1451 PET/CT scan. This scan is done with a radiotracer called 18F-AV1451 (TAU) that will find small areas of tau (abnormal protein) in the brain.
  Other Names: TAU
  Arms: Parametric Imaging
Device: Siemens E7 Reconstruction Tool — Software to correct for motion
  Arms: Motion Correction

SUMMARY:
The purpose of this study is to assess the effectiveness of new software available on a new PET/CT scanner in the Molecular Imaging Research PET/CT Facility. Further, the study aims to evaluate the data acquisition and image processing workflow.

DETAILED DESCRIPTION:
The study will be separated into three cohorts: Motion Correction, Parametric Imaging, and MAP Reconstruction. The motion correction (Aim 1) cohort will involve a group of 30 subjects who are already enrolled in Mayo Clinic Rochester research study 08-005553 (PI: Dr Val Lowe) and are scheduled to be scanned on the Siemens Biograph Vision 600 PET/CT system in the PET/CT Molecular Imaging Research Center in Charlton 6 of Mayo Clinic Rochester. The data gathered from this cohort will assess the effectiveness of motion correction software for patients undergoing PET brain scans. The parametric imaging (Aim 2) cohort will include 30 subjects that have recently undergone a brain or whole body oncologic PET/CT scans on the V600-R1. The purpose of this cohort is to assess the data acquisition and image processing workflow for parametric analysis of brain and whole body scans. The MAP Reconstruction Cohort (Aim 3) is a retrospective study to assess the quality of PET images reconstructed with maximum a posteriori (MAP) reconstruction algorithm.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Subjects who are able and willing to sign the informed consent
* Subjects who are able to follow verbal commands
* A negative urine pregnancy test within 48 hours prior to PET imaging procedures in females of childbearing potential
* Subjects who are scheduled for a PET/CT study under Mayo Clinic Rochester IRB research protocol 08-005553 (Aim 1 cohort only)
* A positive 18F-FDG oncology PET/CT exam in the last six months (Aim 2 cohort only)

Exclusion Criteria:

* Patients who are unable to lay still for an additional 15 minutes (for Aim 1 cohort)
* Patients who are unable to lay still for 90 min for 18F-FDG scans or 100 min for 18F-AV1451 scans (for Aim 2 cohort)
* Patients who cannot follow the prep instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Kemp, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SNMMI abstract on parametric imaging — https://jnm.snmjournals.org/content/62/supplement_1/1412
- See also: SNMMI abstract on brain motion correction — https://jnm.snmjournals.org/content/65/supplement_2/242242

RESULTS

PARTICIPANT FLOW:
Groups:
- Motion Correction: Motion Correction involved the prospective data collection of subjects who were already enrolled in Mayo Clinic Rochester research study 08-005553 (PI: Dr Val Lowe) and were scheduled to be scanned on the Siemens Biograph Vision 600 PET/CT system (hereafter referred to as the V600-R1) in the PET/CT Molecular Imaging Research Center on Charlton 6 of Mayo Clinic Rochester. The purpose of this arm was to evaluate the effectiveness of motion correction software.
  Siemens E7 Reconstruction Tool: Software to correct for motion
- Parametric Imaging: Parametric Imaging involved the prospective data collection of subjects who underwent brain or whole-body oncologic PET/CT scans on the V600-R1. The purpose of this arm was to evaluate the data acquisition and image processing workflow.
  18F-FDG: participants underwent a 18F-FDG PET/CT scan. This scan was done with a radiotracer called 18F-fluorodeoxyglucose (FDG). FDG looks at cellular activity.
  18F-AV1451: participants underwent a 18F-AV1451 PET/CT scan. This scan was done with a radiotracer called 18F-AV1451 (TAU) that finds small areas of tau (abnormal protein) in the brain.
- MAP Reconstruction: MAP reconstruction involved the retrospective data collection of clinically indicated patient scans with the new MAP reconstruction algorithm and compared it to our standard reconstruction algorithm.
Period: Overall Study
Arm/Group | Motion Correction | Parametric Imaging | MAP Reconstruction
Started | 30 | 20 | 30
Completed | 30 | 20 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motion Correction | Parametric Imaging | MAP Reconstruction | Total
Number analyzed (Participants) | 30 | 20 | 30 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 13 | 40
  >=65 years | 16 | 7 | 17 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 14 | 37
  Male | 17 | 10 | 16 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 20 | 28 | 78
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 29 | 20 | 30 | 79
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 20 | 30 | 80

OUTCOME MEASURES:

1. Primary Outcome: Motion Correction
Description: Confirm that motion-corrected reconstructed images acquired when the subject was moving provides similar image quality to the baseline reference reconstructed images acquired when the subject was instructed to remain still. For each subject compute the cumulative absolute relative difference (ARD) histogram in standard uptake values in grey matter voxels in images with and without motion correction versus a reference image for which the subject was stationary, then calculate the percentage of voxels with an ARD greater than 10%. Calculate mean and standard deviation across all subjects. For this measurement 0% is ideal.
Time Frame: 2 years
Population: This outcome measure was collected and analyzed for the Motion Correction arm only.
Measure: Mean (Standard Deviation); unit: percentage of voxels
Arm/Group | Motion Correction
Number analyzed (Participants) | 30
percentage of voxels
  without motion correction | 57.4 (8.5)
  with motion correction | 13.9 (7.4)

2. Primary Outcome: Parametric Imaging
Description: Metabolic rate of 18F-FDG measured from dynamic PET images. Uptake rate constant Ki in the grey matter of the brain.
Time Frame: 2 years
Population: This outcome measure was collected and analyzed for the Parametric Imaging arm only.
Measure: Mean (Standard Deviation); unit: ml/min/ml
Arm/Group | Parametric Imaging
Number analyzed (Participants) | 20
ml/min/ml | 0.0311 (0.0025)

3. Primary Outcome: Map Reconstruction
Description: Confirm that maximum a posteriori reconstructed PET images are diagnostically acceptable. Calculate the Signal-to-Noise ratio (SNR) of the liver and of lesions in images reconstructed with clinical reconstruction (OPTOF) and with MAP (maximum a posteriori) reconstruction. Compute the median and range of SNR for liver and lesions for OPTOF and MAP reconstructions.
Time Frame: 2 years
Population: This outcome measure was collected and analyzed for the MAP reconstruction arm only.
Measure: Median (Full Range); unit: ratio
Arm/Group | MAP Reconstruction
Number analyzed (Participants) | 30
ratio
  SNR in liver for OPTOF | 17 [11 to 29]
  SNR in liver for MAP | 16 [12 to 31]
  SNR in lesions for OPTOF | 37 [10 to 182]
  SNR in lesions for MAP | 48 [14 to 275]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected at baseline, for approximately fifteen minutes.
Arm/Group | Motion Correction | Parametric Imaging | MAP Reconstruction
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/20 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/20 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/20 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT04417998/Prot_000.pdf